CLINICAL TRIAL: NCT06392854
Title: Insulin Regulation of Regional Lipolysis
Brief Title: Regional Lipolysis Insulin Regulation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael D. Jensen, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23-002995; R01DK040484 (NIH)
Record Dates: First submitted 2024-04-24; First posted 2024-05-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: obese vs lean
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- obesity status (Other): obesity
  Interventions: Drug: Insulin
- lean (Other): non-obese
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — 2 dose insulin infusion 4 hours

SUMMARY:
Adults who gain most of their excess weight in the abdominal area typically do not respond to insulin in the same way as lean adults. Researchers are trying to understand why fat tissue responds differently in people with different body types.

DETAILED DESCRIPTION:
Measure regional free fatty acid (FFA) release in volunteers with and without UBO under two different conditions that suppress lipolysis and a condition that markedly stimulates lipolysis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-65years who are able to comprehend instructions, follow study procedures and who willing to provide written, informed consent will be included. The volunteers will consume an isoenergetic diet eating all meals from Mayo Clinical Research Trials Unit (CRTU) for 3 days prior to study.
* Overweight/Obese volunteers will have a BMI 29.0 - 37.0 kg/m2

  * Upper body/visceral obesity (UBO) in women will be defined as those with a waist-hip ratio (WHR) > 0.85 and/or increased visceral fat by single slice CT scan, usually with > 120 cm2 of visceral fat by CT scanning or a visceral fat/total fat ratio of > 0.30, and/or biochemical evidence of metabolic syndrome as defined by ATP III criteria (fasting plasma triglycerides ≥ 150 mg/dL, HDL-cholesterol < 50 mg/dL for women and < 40 mg/dL for men, fasting plasma glucose ≥ 100 mg/dL). Upper body obesity in men will be defined as a waist-hip ratio of >0.95 and/or increased visceral fat (visceral fat area > 180 cm2 or a visceral/total fat abdominal ratio by CT of > 0.40) by single slice CT scan and/or biochemical evidence of metabolic syndrome as defined by adenosine triphosphate (ATP) III criteria. These visceral fat values are based upon the data collected at Mayo Clinic using our methods, and are correlated with dyslipidemia and hyperinsulinemia.
  * Lower body obesity (LBO) in women will be defined as a waist-hip ratio of <0.75 and/or a lower visceral fat by single slice CT scan, usually < 120 cm2 or a visceral fat/total fat ratio of ≤ 0.30 and fasting plasma triglycerides within the normal range. The term "lower body men" is used to describe a male phenotype that is characteristic of adipose insulin sensitivity even with excess body fat. A waist to hip ratio isn't suitable for this description as it is for women. LBO men will be defined as obese men with normal fasting plasma triglycerides, normal fasting plasma glucose and greater proportional leg fat via dual-energy x-ray absorptiometry (DEXA).
* Female subjects are eligible if they meet the following criteria:

  * Are not pregnant or nursing.
  * All women of childbearing potential will have a negative urine pregnancy test at screening and a negative urine pregnancy test day of admission for inpatient study visit.

Exclusion Criteria:

* Individuals with a history of a disease process such as:

  * Ischemic heart disease
  * Atherosclerotic valvular disease
  * Persistent blood pressure greater than 160/95 despite antihypertensive medication
* Smokers
* Diagnosis Diabetes Mellitus
* Concomitant use of medications that can alter free fatty acid metabolism, including, but not limited to niacin, thiazolidinediones, beta-blockers, oral or injected corticosteroids or anabolic steroids.
* Allergy to lidocaine
* Allergy to indocyanine green.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
palmitate release | The study will be conducted in a single day and will last approximately 6 hours
  regional palmitate release rates (micromol/min) will be measured using a combination of leg and splanchnic blood flow combined with stable isotope tracer measurements of palmitate uptake and release across the leg and splanchnic bed. Upper body, non-splanchnic palmitate release will be calculated as: total palmitate release - (splanchnic palmitate release + (leg palmitate release x 2)). Release rates will be measured at baseline (overnight fasting) and in response to the infusion of insulin at low and medium rates. This will allow us to create dose-response curves for leg, splanchnic and upper body non-splanchnic adipose tissue palmitate release.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jensen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No